CLINICAL TRIAL: NCT02441257
Title: Incidence of Gastroesophageal Reflux During LMA Application in Control and Spontaneous Ventilation
Brief Title: Gastroesophageal Reflux During LMA in Control Ventilation (LMA, Laryngeal Mask Airway)
Acronym: LMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhenmeng Wang (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Zhenmeng Wang, Doctor, Eastern Hepatobiliary Surgery Hospital
Organization: Eastern Hepatobiliary Surgery Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: EHBH
Record Dates: First submitted 2015-01-25; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux; Laryngeal Mask Airway; Control Ventilation; Spontaneous Ventilation
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- control ventilation (Experimental): patients are scheduled to receive control or spontaneous ventilation
  Interventions: Procedure: control ventilation; Procedure: spontaneous ventilation

INTERVENTIONS:
Procedure: control ventilation — patients are randomly divided to receive control or spontaneous ventilation randomly.
Procedure: spontaneous ventilation — patients are randomly divided to receive control or spontaneous ventilation randomly.

SUMMARY:
Laryngeal mask airway is seldom used for control ventilation in America, while it is popular in China. The question is whether the incidence of gastroesophageal reflux in control ventilation is really higher than in spontaneous ventilation. So the investigators combine the third generation laryngeal mask and catheter-based Digitrapper ph-Z monitor system to evaluate the exact incidence of gastroesophageal reflux in these two groups.

DETAILED DESCRIPTION:
Patients scheduled for LMA ventilation are divided into two groups randomly, control ventilation group and spontaneous ventilation group. After the third generation laryngeal mask is inserted, catheter-based Digitrapper ph-Z monitor system is applied to measure the exact incidence of gastroesophageal reflux in these two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients for lower extremity operations;
* patients for urological operations;
* patients for gynecological operations.

Exclusion Criteria:

* gastroesophageal reflux disease;
* body mass index more than 30.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
incidence of gastroesophageal reflux of participants | participants will be monitored for the duration of laryngeal mask application, an expected average of 1.5 hours
  evaluate the exact incidence of reflux in LMA patients with catheter-based Digitrapper ph-Z monitor system

CONTACTS AND LOCATIONS:
Overall Officials: Zhenmeng Wang, Doctor, Principal Investigator — Eastern Hepatobiliary Surgery Hospital